CLINICAL TRIAL: NCT05855538
Title: Machine Learning and Artificial Intelligence for Early Detection of Stroke and Atrial Fibrillation. Clinical Cohorts for Validation of New Digital Biomarkers
Brief Title: Clinical Cohorts for Validation of New Digital Biomarkers
Acronym: MAESTRIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Atrial Fibrillation Network (Other)
Responsible Party: Sponsor
Other Study IDs: MAESTRIA-AFNET10
Record Dates: First submitted 2023-03-20; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — optional extra blood for MAESTRIA Biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Paroxysmal AF: 200 patients
- Persistent AF: 200 patients
- Permanent AF: 200 patients

SUMMARY:
The MAESTRIA study is an international, multi-centre, non-interventional, observational registry. The main goal is to enrol a representative group of European patients diagnosed with Atrial Fibrillation (AF) to analyse clinical and relevant parameters (digitalised ECG, echocardiograms, cardiac CTs, MRIs and blood biomarkers) that could be used during clinical practise for the diagnosis of atrial cardiomyopathy. The AF patients will be distributed in 3 groups according to the different manifestation of AF: paroxysmal, persistent and permanent AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and stroke are major health care problems in Europe. They are most often the clinical expression of atrial cardiomyopathy, which is under-recognised due to the lack of specific diagnostic tools. Multidisciplinary research and stratified approaches are urgently needed to prevent, diagnose, and treat AF and stroke and preempt the AF-related threat to healthy ageing in Europe.

MAESTRIA is a European consortium of 18 clinicians, scientists and pharma industry partners who are at the forefront of research and medical care of AF and stroke patients funded by the EU Horizon 2020 programme (grant number 965286). The Atrial Fibrillation Network (AFNET) is one of the 18 partner institutions in this European consortium.

MAESTRIA will create multi-parametric digital tools based on a new generation of biomarkers that integrate artificial intelligence (AI) processing and big data from cutting edge imaging, electrocardiography and omics technologies. It will develop novel biomarkers, diagnostic tools and personalized therapies for atrial cardiomyopathy.

The MAESTRIA-AFNET 10 Study is an integral part of the MAESTRIA project. The study will collect relevant clinical parameters for AF from patients, this includes ECGs, cardiac CTs, MRIs and echocardiograms. Dedicated core labs will collect and homogenize the clinical data.

For atrial arrhythmias (AA) and vascular stiffness index (VSI) recording, patients will be provided with a measuring bracelet for continuous monitoring of heart rhythm with a photoplethysmographic (PPG) sensor coupled with a smartphone app and the Preventicus Heartbeats® analytic service (Class IIa, CE marked), approved as consumer device. Preventicus is ISO 13485 certified.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal AF, persistent AF or permanent AF.
* Patients (or legally acceptable representative if applicable to country specific regulations) provide written informed consent to participate in the study. The patient has the option to give separate consent to donate extra volume of blood during the routine blood collection, that can be used for biomedical research.
* Patient is at least 18 years old.
* Patient must own a smartphone with Apple iOS version 14.5 (or higher) or with Android version 8.0 (or higher).

Exclusion Criteria:

* Any disease that limits life expectancy to less than 1 year.
* All persons unable to provide informed consent.
* All persons exempt from participation in a study or trial by law.
* Any medical or psychiatric condition which, in the investigator´s opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: European prospective cohort of patients with diagnosed AF.
  Patients are distributed in 3 groups according to the different clinical manifestation of AF:
  1. Patients with paroxysmal AF (clinically defined as AF episodes less than one week), or
  2. Patients with persistent AF (clinically defined as AF episodes longer than one week), or
  3. Patients with permanent AF (no documented sinus rhythm or possibility to restore sinus rhythm by any means)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Physical examination | 12 months
  Weight (Kilograms-Kg) Height (centimeters-cm) Weight and height will be combined to calculate BMI in Kg/m^2
Clinically relevant changes in CT/MRI | 12 months
  only if clinically indicated
Atrial Arrythmias (AA) burden and vascular stiffness (measured by a measuring bracelet) | 12 months
  AA burden and vascular stiffness measured by the measuring bracelet
Cognitive function test (MoCA) | Baseline and Follow up at 12 months
  evaluation of cognitive function (includes different tasks: visual/executive; naming; memory; attention; language; abstraction; delayed recall; orientation). Total score will be calculated and collected.
EQ-5D-5L Quality of Life questionnaire | Baseline and Follow up at 12 months
  quality of life assessment (includes questions about mobility, self care, usual activities, pain/discomfort and anxiety/depression). The health state code will be collected (calculated as concatenation of 5 scores). Health score from vertical visual analogue scale (0-100) will be collected.
Ischaemic events (systemic, myocardial and cerebral) | 12 months
  ischaemic events
Echo analysis (TEE_transesophageal echocardiography): LAA smoke available | 12 months
  collected as Yes/No
Echo analysis (TEE_transesophageal echocardiography): Flow velocity in LAA | 12 months
  measured in cm/sec
Echo analysis (TEE_transesophageal echocardiography): Antrum diameter | 12 months
  measured in mm
Echo analysis (TTE_transthoracic echocardiography): LVEF | 12 months
  Measured in %; Biplane Simpson Method
Echo analysis (TTE_transthoracic echocardiography): LA diameter | 12 months
  measured in mm
  LA volume (mL) Septum thickness (mm) Degree of mitral valve insufficiency (Grade I/trivial; Grade II/moderate; Grade III/moderate to severe; Grade IV/severe; None).
  Degree of tricuspid valve insufficiency (Grade I/trivial; Grade II/moderate; Grade III/moderate to severe; Grade IV/severe; None).
Echo analysis (TTE_transthoracic echocardiography): LA volume | 12 months
  measured in mL
Echo analysis (TTE_transthoracic echocardiography): Septum thickness | 12 months
  measured in mm
  Degree of mitral valve insufficiency (Grade I/trivial; Grade II/moderate; Grade III/moderate to severe; Grade IV/severe; None).
  Degree of tricuspid valve insufficiency (Grade I/trivial; Grade II/moderate; Grade III/moderate to severe; Grade IV/severe; None).
Echo analysis (TTE_transthoracic echocardiography): Degree of mitral valve insufficiency | 12 months
  Grade I/trivial; Grade II/moderate; Grade III/moderate to severe; Grade IV/severe; None
Echo analysis (TTE_transthoracic echocardiography): Degree of tricuspid valve insufficiency | 12 months
  Grade I/trivial; Grade II/moderate; Grade III/moderate to severe; Grade IV/severe; None
ECG analysis | 12 months
  Electrocardiogram analysis (paper and digital, if available).
  - 12-lead body surface ECG will be collected.
  Variables to be collected in the eCRF:
  Heart Rhythm (Sinus rhythm; Atrial Fibrillation; Continuous pacing; Pacing and AF; other (specify as free text).
  Heart rate (beats/min) Heart axis (degrees) QRS interval (msec) PR interval (msec) P-wave duration (msec) QT-duration (msec) QTcF (msec) Other relevant ECG findings (to add as free text).
MRI analysis: LAEF | 12 months
  Left atrial ejection fractio measured in %
MRI analysis: LAVi | 12 months
  LAVi left atrial volume index measured in ml/m^2
MRI analysis: LALRS | 12 months
  LALRS left atrial longitudinal reservoir strain measured in %
MRI analysis: LALBS | 12 months
  LALBS left atrial longitudinal booster strain measured in %
CT scan analysis | 12 months
  The cardiac CTs will be sent to the specialised core lab for analysis.
  The analysis will include:
  Atriomic risk of stroke (5 year event risk) Yes/No

SECONDARY OUTCOMES:
CT scan: Atriomic risk for AF | 12 months
  5 year event risk: Yes/No
CT scan: Epicardial Adipose tissue volume | 12 months
  measured in cm^3
CT scan: Epicardial adipose tissue mean attenuation | 12 months
  measured in HU
CT scan: Left atrium volume | 12 months
  measured in cm^3

CONTACTS AND LOCATIONS:
Overall Officials: Stéphan Hatem, Prof, Study Director — ICAN Nutrition Education and Research
Locations (1):
- St Vincenz Hospital, Paderborn, Germany